CLINICAL TRIAL: NCT04513964
Title: Impact of COVID-19 on the Benefit of Cardiac Rehabilitation
Acronym: REACARDIOCOVID
Status: Withdrawn | Type: Observational
Why Stopped: The project was abandoned.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: READCARDIOCOVID
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; Covid19
MeSH Terms: conditions — Heart Failure; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patient not suffering from COVID-19
- COVID-19: Patient who has been infected with COVID-19 with suggestive signs and authentication by PCR or thoracic CT or serology

SUMMARY:
The COVID-19 attack is polymorphic with otorhinolaryngological, pneumological, cardiac, digestive, neurological, muscular attacks with a higher mortality in subjects with comorbidity [> 70 years old, cardiovascular history in particular Arterial hypertension (hypertension ), heart disease…]. This polymorphism is linked to vasculitis and the immune response.

Patients with cardiovascular disease are particularly at risk of decompensating, particularly due to the increased metabolism induced by viral infection and reduced cardiovascular capacities.

On the cardiovascular level, two sides can be considered. On the one hand, cardiovascular disease (hypertension, coronary artery disease) is a comorbid factor. On the other hand, the myocardial damage reflected by the increase in troponin or an alteration of the ejection fraction is a very clear risk factor for death or severe form.

Cardiovascular involvement is particularly high in hospitalized and deceased patients. The odds ratio calculated in a meta-analysis of severe forms of covid-19 with hypertension is 3 [1.9; 3.1], for cardiovascular pathologies of 2.93 [1.73; 4.96]. Recommendations were made for pulmonary rehabilitation but not for cardiovascular rehabilitation.

Cardiac rehabilitation is indicated in most cardiovascular pathologies (after acute coronary syndrome, after coronary angioplasty, in heart failure, after coronary or valve heart surgery, etc.).

It consists of a multidisciplinary approach combining therapeutic pharmacological adjustment, physical activity, therapeutic education in order to improve physical capacities for exertion and reduce morbidity and mortality. The physical exercises can be endurance or resistance type.

Capacity gain at the end of rehabilitation is measured by visual scales, quality of life questionnaires, and a stress test at the start and end of rehabilitation. Most often, rehabilitation centers only do the stress test and estimate through questioning for subjective improvement.

The hypothesis is that patients who contracted COVID-19 would have lower cardiac capacities after recovery from the infection than patients without COVID-19 or that their capacity for recovery would be less. There could be a difference in recovery after cardiac rehabilitation between the two populations regardless of whether the cardiac damage requiring rehabilitation was triggered by COVID-19 or was pre-existing.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient referred for outpatient cardiovascular rehabilitation in one of the participating centers between 02/01/2020 and 12/31/2020
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objecting to the use of their data as part of this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out on the data of patients referred for outpatient cardiovascular rehabilitation in one of the participating centers between 02/01/2020 and 12/31/2020, patients affected or not by COVID-19, i.e. around 60 patients in total.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Impact of COVID-19 on exercise capacity gain after cardiovascular rehabilitation | Month 3
  This outcome corresponds to the difference between the average gain in exercise capacity after cardiac rehabilitation between the two groups of patients Control and COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: DUC Philippe, MD, Study Director — Fondation Hôpital Saint-Joseph

REFERENCES:
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Chen T, Wu D, Chen H, Yan W, Yang D, Chen G, Ma K, Xu D, Yu H, Wang H, Wang T, Guo W, Chen J, Ding C, Zhang X, Huang J, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 26;368:m1091. doi: 10.1136/bmj.m1091. PMID 32217556
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Guan WJ, Liang WH, Zhao Y, Liang HR, Chen ZS, Li YM, Liu XQ, Chen RC, Tang CL, Wang T, Ou CQ, Li L, Chen PY, Sang L, Wang W, Li JF, Li CC, Ou LM, Cheng B, Xiong S, Ni ZY, Xiang J, Hu Y, Liu L, Shan H, Lei CL, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Cheng LL, Ye F, Li SY, Zheng JP, Zhang NF, Zhong NS, He JX; China Medical Treatment Expert Group for COVID-19. Comorbidity and its impact on 1590 patients with COVID-19 in China: a nationwide analysis. Eur Respir J. 2020 May 14;55(5):2000547. doi: 10.1183/13993003.00547-2020. Print 2020 May. PMID 32217650
- [Result] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Result] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362
- [Result] Lippi G, Lavie CJ, Sanchis-Gomar F. Cardiac troponin I in patients with coronavirus disease 2019 (COVID-19): Evidence from a meta-analysis. Prog Cardiovasc Dis. 2020 May-Jun;63(3):390-391. doi: 10.1016/j.pcad.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32169400